CLINICAL TRIAL: NCT00621296
Title: Phase II Study of MP-424 in Patients With (Genotype 1b) Hepatitis C
Brief Title: Safety and Efficacy of MP-424 to Treat Chronic Hepatitis C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Collaborators: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G060-A7
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Results first posted 2012-10-19 (Estimated); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Hepatitis C
Keywords: Chronic Hepatitis C; Protease Inhibitor
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic | interventions — telaprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MP-424 (Experimental)
  Interventions: Drug: MP-424 (Telaprevir)

INTERVENTIONS:
Drug: MP-424 (Telaprevir) — Three tablets of MP-424 250mg tablet at a time, every 8 hours, 24 weeks administration (dose in a day: 2250 mg)
  Other Names: Telaprevir

SUMMARY:
The purpose of this study is to assess the efficacy and safety after administration of MP-424 to patients with chronic hepatitis C.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with genotype 1b chronic hepatitis C
* Patients naive to the concomitant medications with interferon

Exclusion Criteria:

* Patients diagnosed with decompensated cirrhosis
* Patients diagnosed with positive HBs antigen in the test

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-01; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fumitaka Suzuki, MD, Principal Investigator — Department of Hepatology, Toranomon Hospital
Locations (1):
- Toranomon Hospital, Kawasaki, Takatsu-ku, Japan

REFERENCES:
- [Result] Toyota J, Ozeki I, Karino Y, Asahina Y, Izumi N, Takahashi S, Kawakami Y, Chayama K, Kamiya N, Aoki K, Yamada I, Suzuki Y, Suzuki F, Kumada H. Virological response and safety of 24-week telaprevir alone in Japanese patients infected with hepatitis C virus subtype 1b. J Viral Hepat. 2013 Mar;20(3):167-73. doi: 10.1111/j.1365-2893.2012.01640.x. Epub 2012 Jul 13. PMID 23383655

RESULTS

PARTICIPANT FLOW:
Groups:
- MP-424: Drug: MP-424 750 mg every 8 hours for 24 weeks Other Name: Telaprevir
Period: Overall Study
Arm/Group | MP-424
Started | 15
Completed | 1
Not Completed | 14
Not completed — Adverse Event | 2
Not completed — Lack of Efficacy | 1
Not completed — Physician Decision | 7
Not completed — Unmatch Criteria | 1
Not completed — Stopping Criteria | 3

BASELINE CHARACTERISTICS:
Arm/Group | MP-424
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Undetectable HCV RNA at 24 Weeks After Completion of Drug Administration
Time Frame: 24 Weeks After Completion of Drug Administration (dosing period is 24 Weeks) or drug withdrawal. The subjects were assessed at 24 weeks following the last dose of study drug.
Measure: Number; unit: participants
Arm/Group | MP-424
Number analyzed (Participants) | 15
participants | 1

ADVERSE EVENTS:
Arm/Group | MP-424
Serious Adverse Events (participants affected / at risk) | 1/15
Other Adverse Events (participants affected / at risk) | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MP-424 (N=15)
Herpes zoster (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MP-424 (N=15)
Anaemia (Blood and lymphatic system disorders) | 7
Anorexia (Metabolism and nutrition disorders) | 3
Headache (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 8
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Nocturia (Renal and urinary disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 2
Malaise (General disorders) | 1
Thirst (General disorders) | 2
Low density lipoprotein increased (Investigations) | 6
Blood uric acid increased (Investigations) | 4
Blood triglycerides increased (Investigations) | 2
Blood creatinine increased (Investigations) | 2
Blood lactate dehydrogenase increased (Investigations) | 1
Platelet count decreased (Investigations) | 2
Protein urine present (Investigations) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1
Blister (Skin and subcutaneous tissue disorders) | 1
Oedema (General disorders) | 1
Blood urine present (Investigations) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1
Nasopharyngitis (Infections and infestations) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Periodontitis (Gastrointestinal disorders) | 1
White blood cell count decreased (Investigations) | 1
Insomnia (Psychiatric disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other